CLINICAL TRIAL: NCT05206942
Title: Serial Ultrasound of Solid Tumor Lesions to Detect Early Response to Cancer Immunotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-59526; NCI-2022-02835 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program); 5R21CA259756-02 (NIH)
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Ultrasonography, Doppler; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ultrasound (Experimental): Patients receiving standard of care immune checkpoint inhibitor are followed with the ultrasound studies at treatment baseline, 3 weeks and 6 weeks.
  Interventions: Diagnostic Test: Doppler ultrasound; Diagnostic Test: Long Ensemble Angular-coherence Doppler [LEAD] ultrasound; Diagnostic Test: Contrast-enhanced ultrasound (CEUS)

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound — Power Doppler measurements will be made using a portable Siemens S2000 or S3000 ultrasound scanner
Diagnostic Test: Long Ensemble Angular-coherence Doppler [LEAD] ultrasound — Long Ensemble Angular-coherence Doppler measurements will be made using a Verasonics Vantage 256 scanner
Diagnostic Test: Contrast-enhanced ultrasound (CEUS) — Contrast-enhanced ultrasound measurements will be made using Lumason IV contrast injection followed by an injection of normal saline

SUMMARY:
Primary objective is to assess whether changes in quantitative tumor perfusion parameters after 3 weeks of treatment, as measured by CEUS, can predict initial objective response to therapy, defined by current standard-of-care

Secondary objectives are to evaluate if there is an optimal ultrasound imaging modality (CEUS or conventional power Doppler or LEAD ultrasound) or optimal time point to predict initial objective response and to assess the correlation of tumor perfusion parameters with change in overall tumor burden, change in diameter on a per-lesion basis, and with 12-month progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* at least one solid tumor lesion greater than 1 cm in diameter (primary tumor and/or at metastatic site), amenable to ultrasound imaging
* planned to be treated with ICI therapy (single agent or in combination with any other drug)
* written informed consent.

  * prior use of any ICI is not necessarily excluded, and patients may be included with the approval of the Protocol Director

Subjects may participate in the study more than once at the discretion of the Protocol Director, for example, if they receive different lines of treatment that all qualify for the study.

Exclusion Criteria:

* known hypersensitivity to sulfur hexafluoride lipid microsphere or its components, such as polyethylene glycol (PEG)
* any comorbid condition that, in the opinion of the treating provider or the Protocol Directors, compromises the participant's ability to participate in the study

  * Examples: any mental condition that compromises the ability to follow a consent discussion, or to make informed decisions (except if represented by a Legally Authorized Representative [LAR]), or to have ultrasound exams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Initial objective response per RECIST v1.1 | 16 weeks
  Initial objective response is defined as having either Complete Response (CR) or Partial Response (PR) per RECIST v1.1

SECONDARY OUTCOMES:
Initial relative change in tumor burden | 16 weeks
  defined as relative change in the sum of diameters of all measurable tumors, assessed between treatment 'baseline' and first on-treatment response evaluation
Initial lesion response | 16 weeks
  defined as the relative change in tumor diameter of a single lesion between treatment 'baseline' and first on-treatment response evaluation
progression-free survival (PFS) | 12 months
  defined as not having experienced any PD per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Alice C. Fan, MD, Principal Investigator — Stanford University; Jeremy Dahl, Ph.D, Principal Investigator — Stanford University; Aya Kamaya, M.D, Principal Investigator — Stanford University
Locations (1):
- Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No